CLINICAL TRIAL: NCT04734275
Title: A Randomised, Single-dose, Open-label, Single-centre, Crossover Study to Assess the Relative Bioavailability and Safety of Different Formulations of AZD5718 in Fasted and Fed State in Healthy Volunteers
Brief Title: Study to Assess Relative Bioavailability and Safety of AZD5718 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7551C00003
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Disease
Keywords: AZD5718; Bioavailability; 5-lipoxygenase activating protein (FLAP) inhibitor; Safety and tolerability
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — AZD5718

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Test Formulation): AZD5718 Dose A, fasted (Experimental): Subjects will receive single dose of AZD5718 (Dose A), in fasted condition.
  Interventions: Drug: AZD5718
- Treatment B (Test Formulation): AZD5718 Dose A, fed (Experimental): Subjects will receive single dose of AZD5718 (Dose A) in fed condition
  Interventions: Drug: AZD5718
- Treatment C (Reference Formulation): AZD5718 Dose A, fasted (Active Comparator): Subjects will receive single dose of AZD5718 (Dose A) in fasted condition
  Interventions: Drug: AZD5718

INTERVENTIONS:
Drug: AZD5718 — Subjects will receive single doses of AZD5718 on 3 occasions, separated by at least 7 days washout, under fasted and fed conditions.

SUMMARY:
This study will be a randomised, open-label, 3-period, 3-treatment, single-dose, crossover study in healthy subjects The study will be performed at a single study centre in the United Kingdom.

DETAILED DESCRIPTION:
The study will comprise:

* A screening period of maximum 28 days;
* 3 treatment periods during which subjects will be resident at the Clinical Unit from the day before dosing with AZD5718 (Day -1) until at least 48 hours after dosing (Day 3), with discharge on the morning of Day 3 of each treatment period; and
* A final visit within 5 to 7 days after the last administration of AZD5718.

Subjects will receive single doses of AZD5718 on 3 occasions, separated by at least 7 days washout, under fasted and fed conditions. Two different formulations (Test Formulation and Reference Formulation) will be given in a randomised order:

* Treatment A (Test Formulation): AZD5718 Dose A, fasted
* Treatment B (Test Formulation): AZD5718 Dose A, fed
* Treatment C (Reference Formulation): AZD5718 Dose A, fasted

ELIGIBILITY:
Only key inclusion and exclusion criteria are presented here:

Inclusion Criteria:

* Healthy male and/or female subjects aged 18 - 55 years inclusive with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at each admission to the unit, must not be lactating and must be of nonchildbearing potential, confirmed at the Screening Visit.
* Male subjects must adhere to the contraception methods as detailed in protocol.
* Have a body mass index between 18.5 and 30 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the principal investigator (PI), may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational Medicinal Product (IMP).
* Any clinically significant abnormalities in clinical chemistry, haematology, coagulation, or urinalysis results, at the Screening Visit and/or on admission to the Clinical Unit for Treatment Period 1 as judged by the PI including:

  * Alanine aminotransferase > upper limit of normal (ULN)
  * Aspartate aminotransferase > ULN
  * Bilirubin (total) > ULN
  * Gamma glutamyl transferase > ULN
* Any clinically significant abnormal findings in vital signs and 12-lead electrocardiogram at the Screening Visit and/or on each admission to the Clinical Unit, as judged by the Principal Investigator (PI).
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.
* Any positive result on screening for IgM. If positive for IgG, a reverse transcriptase polymerase chain reaction test for severe acute respiratory syndrome coronavirus 2 must be performed on the same day and if positive, the subject is excluded.
* Known or suspected Gilbert's syndrome.
* Known or suspected significant history of drug abuse.
* Has received another new chemical or biological entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study.
* Plasma donation within 1 month of the Screening Visit or any blood donation/loss more than 500 mL during the 3 months prior to the Screening Visit.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to the Screening Visit.
* Positive screen for drugs of abuse or cotinine at the Screening Visit or on each admission to the Clinical Unit.
* Positive screen for alcohol at the Screening Visit or on each admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), hormonal replacement therapy, herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI. Excessive intake of alcohol defined as the regular consumption of more than 24 g (3 units) of alcohol per day for men or 12 g (1.5 units) of alcohol per day for women.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the PI. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (eg, > 5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the Clinical Unit.
* Subjects who have previously received AZD5718.
* Judgement by the PI that the subject should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects with any special dietary restrictions such as subjects who are lactose intolerant or with food allergies.
* Subjects who cannot eat a standard Food and Drug Administration high-fat breakfast.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from zero to infinity (AUCinf) (Treatment A versus Treatment C) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of the Test Formulation in the fasted state (Treatment A) compared to Reference Formulation in the fasted state (Treatment C) using AUCinf will be assessed.
Area under the plasma concentration-time curve from zero to the last quantifiable concentration (AUClast) (Treatment A versus Treatment C) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of the Test Formulation in the fasted state (Treatment A) compared to Reference Formulation in the fasted state (Treatment C) using AUClast will be assessed.
Maximum observed plasma (peak) drug concentration (Cmax) (Treatment A versus Treatment C) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of the Test Formulation in the fasted state (Treatment A) compared to Reference Formulation in the fasted state (Treatment C) using Cmax will be assessed.
Plasma concentration at 24h post-dose (C24) (Treatment A versus Treatment C) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of the Test Formulation in the fasted state (Treatment A) compared to Reference Formulation in the fasted state (Treatment C) using C24 will be assessed.
AUCinf (Treatment B versus Treatment A) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of Treatment B (fed state, Test Formulation) versus Treatment A (fasted state, Test Formulation) using AUCinf will be assessed.
AUClast (Treatment B versus Treatment A) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of Treatment B (fed state, Test Formulation) versus Treatment A (fasted state, Test Formulation) using AUClast will be assessed.
C24 (Treatment B versus Treatment A) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of Treatment B (fed state, Test Formulation) versus Treatment A (fasted state, Test Formulation) using C24 will be assessed.
Cmax (Treatment B versus Treatment A) | Days 1, 2 and 3 of each Treatment Period (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours)
  Relative bioavailability (Frel) of Treatment B (fed state, Test Formulation) versus Treatment A (fasted state, Test Formulation) using Cmax will be assessed.

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs) and serious AEs | From screening (SAEs only) until Follow-up Visit (5 to 7 days post final dose)
  Safety and tolerability of single doses of AZD5718 in healthy subjects will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, Dr, Principal Investigator — Parexel Early Phase Clinical Unit London, Level 7, Northwick Park Hospital Watford Road, Harrow Middlesex HA1 3UJ UK
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home